CLINICAL TRIAL: NCT00540384
Title: A Randomised, Double-blind, Placebo-controlled, Dose-finding Study of Novel Erythropoiesis Stimulating Protein (NESP) Administered by Subcutaneous (SC) Injection for the Treatment of Anaemia in Subjects With Solid Tumours Receiving Multicycle Chemotherapy
Brief Title: Dose-finding Study of Novel Erythropoiesis Stimulating Protein (NESP) for the Treatment of Anaemia in Subjects With Solid Tumours Receiving Multicycle Chemotherapy
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 980291
Record Dates: First submitted 2007-10-04; First posted 2007-10-08 (Estimated); Last update posted 2013-05-08 (Estimated); Status verified 2013-05

CONDITIONS: Anemia; Solid Tumors
Keywords: Anemia; Solid tumors; Multicycle chemotherapy; NESP
MeSH Terms: conditions — Anemia | interventions — Darbepoetin alfa

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (6):
- NESP - Schedule 1 Part A (Experimental): Part A - 4.5, 6.75, 9.0 or 13.5 mcg/kg Q3W for 12 weeks
  Interventions: Drug: Novel Erythropoiesis Stimulating Protein (NESP) (darbepoetin alfa)
- NESP - Schedule 2 Part A (Experimental): NESP 9.0, 12.0, 15.0 or 18.0 mcg/kg Q4W for 12 weeks
  Interventions: Drug: Novel Erythropoiesis Stimulating Protein (NESP) (darbepoetin alfa)
- Placebo - Schedule 1 Part A (Placebo Comparator): Placebo Q3W for 12 weeks
  Interventions: Drug: Placebo
- NESP - Schedule 1 Part B (Experimental): Open-label NESP at the dose of study drug administered at the end of Part A. Increase dose at week 19 if hgb < 13.0g/dL and/or RBC transfusion in previous 2 weeks.
  Interventions: Drug: Novel Erythropoiesis Stimulating Protein (NESP) (darbepoetin alfa)
- Placebo - Schedule 2 Part A (Placebo Comparator): Placebo Q4W for 12 weeks
  Interventions: Drug: Placebo
- NESP - Schedule 2 Part B (Experimental): Open-label NESP at the dose of study drug administered at the end of Part A
  Interventions: Drug: Novel Erythropoiesis Stimulating Protein (NESP) (darbepoetin alfa)

INTERVENTIONS:
Drug: Placebo — Placebo
  Arms: Placebo - Schedule 1 Part A; Placebo - Schedule 2 Part A
Drug: Novel Erythropoiesis Stimulating Protein (NESP) (darbepoetin alfa) — Novel Erythropoiesis Stimulating Protein (NESP) (darbepoetin alfa)
  Arms: NESP - Schedule 1 Part A; NESP - Schedule 1 Part B; NESP - Schedule 2 Part A; NESP - Schedule 2 Part B

SUMMARY:
The purpose of this study is to assess the safety of NESP administered by SC injection in subjects with solid tumours and anaemia receiving multicycle chemotherapy.

Subjects in this study enter one of two schedules: Schedule 1 or Schedule 2. Schedule 1 is a sequential dose escalation study which consists of Parts A and B. Part A is the initial treatment phase, where the clinically effective dose (CED) of NESP administered every 3 weeks will be determined after 12 weeks of treatment. Part B is an optional 12-week, open-label, dose-maintenance phase that follows Part A.

Schedule 2 is a parallel dose-finding study and also consists of Parts A and B. Part A is the initial treatment phase, where the CED of NESP administered every 4 weeks will be determined after 12 weeks of treatment. Part B is an optional 12-week, open-label, dose-maintenance phase that follows Part A.

ELIGIBILITY:
Inclusion Criteria:

* Subject with solid tumour(s)
* Anaemia (hgb less than or equal to 11.0 g/dL
* Planned to receive cyclic chemotherapy
* At least 6-month life expectancy
* Eastern Cooperative Oncology Group (ECOG) status of 0 to 2
* Adequate renal and liver function
* At least 18 years of age

Exclusion Criteria:

* Central nervous system disease
* Iron deficiency
* Received more than 2 RBC transfusions within 4 weeks before randomisation or any RBC transfusion within 2 weeks before randomisation
* Received recombinant human erythropoietin (rHuEPO) therapy within 8 weeks before randomisation
* History of any seizure disorder
* Cardiac disease
* Active infection or inflammatory disease
* Known positive test for HIV infection
* Known primary haematologic disorder which could cause anaemia
* Use of other investigational agent(s)/device(s)
* Pregnant or breast feeding
* Known hypersensitivity to any recombinant mammalian derived product

Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 405 (Estimated)
Dates: Start 1999-07; Primary Completion 2002-03 (Actual); Study Completion 2002-06 (Actual)

PRIMARY OUTCOMES:
Occurence of adverse events and antibody formation to NESP | throughout the study

SECONDARY OUTCOMES:
Number and proportion of subjects who receive any RBC transfusion, number of units of RBC transfused, and number of days with at least one RBC transfusion during weeks 1-12, 1-4, 5-8, 9-12, and 5-12, with emphasis on the 5-12 week window | during weeks 1-12, 1-4, 5-8, 9-12, and 5-12
Selected domains of quality of life (QOL) measured by FACT-G and FACT-anaemia scales, BSI depression and BSI anxiety scales, and de novo questions | throughout the study
Relationship between these QOL measurements and hgb
Hgb correction to greater than or equal to 12.0 g/dL in the absence of a red blood cell (RBC) transfusion during the preceding 4 weeks during treatment phase | during treatment phase
Number and proportion of subjects, during the treatment phase, who achieve a hemoglobin (hgb) response | during the treatment phase
Time to hgb response and hgb correction after the initiation of treatment | after the initiation of treatment
Change in hgb measured at the end of the treatment phase compared to baseline | baseline to end of the treatment phase

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Result] Kotasek D, Steger G, Faught W, Underhill C, Poulsen E, Colowick AB, Rossi G, Mackey J; Aranesp 980291 Study Group. Darbepoetin alfa administered every 3 weeks alleviates anaemia in patients with solid tumours receiving chemotherapy; results of a double-blind, placebo-controlled, randomised study. Eur J Cancer. 2003 Sep;39(14):2026-34. doi: 10.1016/s0959-8049(03)00456-8. PMID 12957457
- See also: Notice regarding posted summaries of trial results — http://download.veritasmedicine.com/REGFILES/amgen/Amgen_results_disclaimer.pdf
- See also: To access clinical trial results information click on this link — http://download.veritasmedicine.com/REGFILES/amgen/08D_FDAMA_113_Posting_Summary_33_NESP_980291.pdf
- See also: FDA-approved Drug Labeling — http://www.aranesp.com/
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com